CLINICAL TRIAL: NCT03615144
Title: A Phase II Trial of Alpha Beta T-cell and CD19 B-cell Depleted Peripheral Blood Stem Cell Transplantation Using the CliniMACS System for Patients With Non-Malignant Hematologic Disorders From Matched or Mismatched, Related or Unrelated Donors
Brief Title: TCR Alpha Beta T-cell and CD19 B-cell Depleted Peripheral Blood Stem Cell Transplantation Using the CliniMACS System for Patients With Non-Malignant Hematologic Disorders From Matched or Mismatched, Related or Unrelated Donors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Participant accrual low and the study was closed
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-596
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2020-11

CONDITIONS: Non-Malignant Hematologic Disorders
Keywords: T-cell; B-cell; CliniMACS System; Melphalan; Thiotepa; Clofarabine; Fludarabine; 17-596
MeSH Terms: interventions — Melphalan; Thiotepa; Clofarabine; fludarabine; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Intervention Model Description: For this trial, patients will be assigned to receive one of two conditioning regimens, based on their disease, disease severity, organ status and history of red blood cell alloimmunization.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melphalan/Thiotepa/Clofarabine (Active Comparator): Melphalan 70 mg/m2/day x 2, Thiotepa 7.5 mg/kg/day x 2 and Clofarabine 20-30 mg/m2/day x 5. Patients will also receive rabbit anti-thymocyte globulin at 2.5 mg/kg/day x 3 doses prior to the start of conditioning.
  Interventions: Drug: Melphalan; Drug: Thiotepa; Drug: Clofarabine; Drug: Anti-Thymocyte Globulin (Rabbit) (Thymoglobulin®); Procedure: CliniMACS reagents
- Melphalan/Thiotepa/ Fludarabine (Active Comparator): Melphalan 70 mg/m2/day x 2, Thiotepa 7.5 mg/kg/day x 2 and Fludarabine 30 mg/m2/day x 5. Patients will also receive rabbit anti-thymocyte globulin at 2.5 mg/kg/day x 3 doses prior to the start of conditioning.
  Interventions: Drug: Melphalan; Drug: Thiotepa; Drug: Fludarabine; Drug: Anti-Thymocyte Globulin (Rabbit) (Thymoglobulin®); Procedure: CliniMACS reagents

INTERVENTIONS:
Drug: Melphalan — Melphalan 70 mg/m2/day x 2
Drug: Thiotepa — Thiotepa 7.5 mg/kg/day x 2
Drug: Clofarabine — Clofarabine 20-30 mg/m2/day x 5
  Arms: Melphalan/Thiotepa/Clofarabine
Drug: Fludarabine — Fludarabine 30 mg/m2/day x 5
  Arms: Melphalan/Thiotepa/ Fludarabine
Drug: Anti-Thymocyte Globulin (Rabbit) (Thymoglobulin®) — antithymocyte globulin (ATG) (rabbit ATG 2.5 mg/kg/day x 3 or equine ATG 15 mg/kg/day x 3 (or 40 mg/kg/day x 1 equine ATG if rabbit ATG is not tolerated) during pre-transplant conditioning to deplete host T-cells that could hamper engraftment.
Procedure: CliniMACS reagents — Products will then undergo TCR-αβ+ and CD-19 depletion using the CliniMACS.

SUMMARY:
The purpose of this study is to find out if removing a specific type of white blood cell (called alpha beta T-cell) that help make up the transplant donor's stem cells can improve results of blood stem cell transplant for the participant's disease.

ELIGIBILITY:
Subject Inclusion Criteria:

* Lethal disorders of Hematopoiesis correctable by transplant for which Alpha βeta T-cell and CD-19 depleted allogeneic hematopoietic stem cell transplantation is indicated including:
* Sickle cell disease (HbSS, HbSC, HbSB0 thalassemia, HbSB+, HbSD, HbSE) with at least one of the following criteria (Walters et al):

  1. Cerebrovascular accident lasting longer than 24 hours
  2. Impaired neuropsychological function with abnormal brain MRI/MRA
  3. Recurrent hospitalizations (>2 episodes/year over several years) or exchange transfusions for acute chest syndrome
  4. Recurrent priapism
  5. Stage I or II sickle chronic lung disease
  6. Sickle cell nephropathy (moderate to severe proteinuria or glomerular filtration rate 30-50% of predicted normal value for age)
  7. Bilateral proliferative retinopathy with major visual impairment in at least one eye
  8. Osteonecrosis of multiple joints
  9. Red cell alloimmunization during chronic transfusion therapy
* Thalassemia major with at least one of the following criteria:

  1. Age <16 years
  2. Available HLA-identical sibling
  3. Red blood cell transfusion dependency
  4. Lucarelli class 1 or 2 risk status (i.e. with only 0-2 of the following factors: hepatomegaly, portal fibrosis, or poor response to chelation therapy)
  5. Recurrence of disease after previous stem cell transplant
* Bone Marrow Failure Syndromes:

  1. Aplastic anemia refractory to immunosuppressive therapy
  2. Diamond Blackfan Anemia refractory to conventional therapy
  3. Shwachman-Diamond Syndrome
  4. Severe Congenital Neutropenia
  5. Congenital Amegakaryocytic Thrombocytopenia
  6. Thrombocytopenia Absent Radii syndrome
  7. Other marrow failure disorders not otherwise specified
* Autoimmune cytopenias refractory to all conventional treatments

  1. Autoimmune hemolytic anemia
  2. Immune thrombocytopenia
  3. Evan's syndrome
  4. Pure red cell aplasia
* Histiocytic disorders:

  1. Hemophagocytic lymphohistiocytosis
  2. High risk, recurrent or refractory Langerhans cell histiocytosis
  3. Secondary HLH

Subject Inclusion Criteria:

* Recipient's age birth to < 70 years old
* Patients must have adequate organ function measured by:
* Cardiac: asymptomatic or if symptomatic then LVEF at rest must be ≥ 50% and must improve with exercise.
* Hepatic: < 3x ULN AST and ≤ 1.5 mg/dl total serum bilirubin, unless there is congenital benign hyperbilirubinemia or if the hyperbilirubinemia is directly caused by the disease in which the patient is receiving a transplant for. Patients with higher bilirubin levels due to causes other than active liver disease are also eligible with PI approval e.g. patients with PNH, Gilbert"s disease or other hemolytic disorders.
* Pulmonary: asymptomatic or if symptomatic, DLCO ≥ 50% of predicted (corrected for hemoglobin).
* Renal: serum creatinine ≤1.5x normal for age. If serum creatinine is outside the normal range, then CrCl > 70 mL/min/1.73m2 (calculated or estimated) or GFR (mL/min/1.72m2) >30% of predicted normal for age.
* Normal GFR in Children and Young Adults.

Donor Inclusion Criteria:

* Each donor must meet criteria outlined by institutional guidelines and be medically eligible to donate according to NMDP (or equivalent donor search organization) criteria including testing for antibodies to Human TLymphotrophic Virus Types I & II (Anti-HTLV-I/II) and screening for West Nile Virus, Creutzfeldt-Jakob disease and Zika.
* Pediatric donors should weigh ≥ 25.0 kg, have adequate peripheral venous catheter access for leukapheresis or must agree to placement of a central catheter.
* Donor should be healthy and agree to receive G-CSF followed by donation of peripheral blood stem cells.
* Donors must agree to anesthesia and marrow donation (in cases of inadequate PBSC collection).
* Related or unrelated donors who are 7/8 or 8/8 HLA-antigen matched for haplotypes A, B, C, DRB1 OR Related donors who are 4-6/8 HLA-antigen matched.

Subject Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Active viral, bacterial or fungal infection
* Patient seropositive for HIV-I/II; HTLV-I/II
* Karnofsky (adult)/Lansky (pediatric) < 70%
* Inherited DNA repair deficiency: Fanconi Anemia and Dyskeratosis Congenita. These are presently undergoing transplantation based on a multi-center protocol
* Patients with Thalassemia major with Pesaro risk score >II
* Inherited metabolic disorders: Hurler Syndrome, Sly syndrome (MPSVIII), α-Mannosidosis, X- ALD, Osteopetrosis

Donor Exclusion Criteria:

* Donors who are seropositive for HIV-I/II or HTLV-I/II and female patients who are pregnant or breastfeeding will not be eligible for this study.

Ages: 1 Year to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cancio, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial SloanKettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Melphalan/Thiotepa/Clofarabine | Melphalan/Thiotepa/ Fludarabine
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Participant no longer eligible for this protocol | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participant accrual low and the study was closed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Melphalan/Thiotepa/Clofarabine | Melphalan/Thiotepa/ Fludarabine | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 20 [20 to 20] |  | 20 [20 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as time from transplant to death or last follow-up. Rate greater than 0.75 would be considered a success.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Melphalan/Thiotepa/Clofarabine | Melphalan/Thiotepa/ Fludarabine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only 1 participants was accrued before the study was closed to accrual due to low accrual
Arm/Group | Melphalan/Thiotepa/Clofarabine | Melphalan/Thiotepa/ Fludarabine
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melphalan/Thiotepa/Clofarabine (N=1) | Melphalan/Thiotepa/ Fludarabine (N=0)
Blood and lymphatic system disorders - Other, spec (Blood and lymphatic system disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT03615144/Prot_SAP_000.pdf